CLINICAL TRIAL: NCT01143545
Title: Allogeneic Tumor Cell Vaccine With Metronomic Oral Cyclophosphamide and Celecoxib as Adjuvant Therapy for Lung and Esophageal Cancers, Thymic Neoplasms, Thoracic Sarcomas, and Malignant Pleural Mesotheliomas
Brief Title: Pilot Study of Allogeneic Tumor Cell Vaccine With Metronomic Oral Cyclophosphamide and Celecoxib in Patients Undergoing Resection of Lung and Esophageal Cancers, Thymic Neoplasms, and Malignant Pleural Mesotheliomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed accrual due to unpromising results and the opening of study 14C0053 targeting the same population.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100138; 10-C-0138
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer; Esophageal Cancer; Malignant Pleural Mesothelioma; Sarcoma; Thymic Carcinoma
Keywords: Cancer Vaccine; Immunotherapy; Adjuvant Therapy; Surgical Intervention; Lung Cancer; Esophageal Cancer; Thymic Carcinoma; Malignant Pleural Mesothelioma
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms; Mesothelioma, Malignant; Sarcoma; Thymoma | interventions — Celecoxib; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Allogeneic tumor cell vaccine + chemotherapy
  Interventions: Biological: Allogeneic Tumor Cell Vaccine (K562); Drug: Celecoxib; Drug: cyclophosphamide

INTERVENTIONS:
Biological: Allogeneic Tumor Cell Vaccine (K562) — Subcutaneous injection monthly for 6 months
Drug: Celecoxib — 400 g po bid
Drug: cyclophosphamide — 50 mg po bid

SUMMARY:
Background:

- Certain types of lung, esophageal, or thymic cancers and mesotheliomas have specific antigens (protein molecules) on their surfaces. Research studies have shown that giving a vaccine that contains antigens similar to these may cause an immune response, which may keep tumors from growing. Researchers are also interested in determining whether the chemotherapy drug cyclophosphamide and the anti-inflammatory drug celecoxib may help the vaccine work better, particularly in patients with lung cancer.

Objectives:

- To evaluate the safety and effectiveness of tumor cell vaccines in combination with cyclophosphamide and celecoxib in patients with cancers involving the chest.

Eligibility:

- Individuals at least 18 years of age who have had surgery for small cell or non-small cell lung cancer, esophageal cancer, thymoma or thymic carcinoma, and malignant pleural mesothelioma.

Design:

* Following recovery from surgery, chemotherapy, or radiation, participants will have leukapheresis to collect lymphocytes (white blood cells) for testing.
* Participants will receive celecoxib and cyclophosphamide to take twice a day at home, 7 days before the vaccine.
* Participants will have the vaccine in the clinical center (one or two shots per month for 6 months), and will stay in the clinic for about 4 hours after the vaccine. Participants will keep a diary at home of any side effects from the vaccine, and will continue to take cyclophosphamide and celecoxib.
* One month after the sixth vaccine, participants will provide another blood sample for testing, and if the tests are satisfactory will return to the clinic every 3 months for 2 additional vaccines.
* Participants will return to clinic for follow-up physical examinations, lab tests, and scans every 3 months for 2 years and then every 6 months for up to 3 years.

DETAILED DESCRIPTION:
Background:

During recent years, the cancer-testis (CT) antigens have emerged as attractive targets for cancer immunotherapy. Whereas lung and esophageal cancers, as well as malignant pleural mesotheliomas express a variety of CT antigens, immune responses to these antigens appear uncommon in patients with these malignancies, possibly due to low-level, heterogeneous antigen expression, as well as immunosuppressive regulatory T cells. Our published studies indicate that numerous CT antigens can be induced in tumor cells by DNA demethylating agents and histone deacetylase (HDAC) inhibitors. Conceivably, vaccination of cancer patients with allogeneic tumor cells expressing high levels of multiple CT antigens in combination with depletion of T regulatory cells will induce broad immunity to these antigens. In order to examine this issue, patients with lung and esophageal cancers, thymic neoplasms, primary thoracic sarcomas, and malignant pleural mesotheliomas will be vaccinated with irradiated K562 erythroleukemia cells expressing GM-CSF (K562-GM) following completion of appropriate combined modality therapy. Vaccines will be administered in conjunction with metronomic oral cyclophosphamide (50 mg PO BID x 7dq 14d), and celecoxib (400 mg PO BID). Serologic responses to a variety of recombinant CT antigens as well as cell-mediated recognition of autologous tumor cells and EBVtransformed B cells will be assessed before and after vaccination.

Objective:

-To assess the safety of K562-GM allogeneic tumor cell vaccines in combination with oral metronomic cyclophosphamide and celecoxib in thoracic oncology patients.

Eligibility:

* Patients with histologically or cytologically proven small cell or non-small cell lung cancer, esophageal cancer, thymoma or thymic carcinoma, primary thoracic sarcomas, and malignant pleural mesothelioma with no evidence of disease (NED) or minimal residual disease (MRD) in the primary site following standard multimodality therapy.
* Patients must be 18 years or older with an ECOG performance status of 0 - 2, without evidence of unstable or decompensated myocardial disease. Patients must have adequate pulmonary reserve evidenced by FEV1 and DLCO equal to or greater than 30% predicted; pCO2 less than 50 mm Hg and pO2 greater than 60 mm Hg on room air ABG; and be on no immunosuppressive medications except inhaled corticosteroids at the time vaccination commences.
* Patients must have a platelet count greater than 100,000, an ANC equal to or greater than 1500 without transfusion or cytokine support, a normal PT, and adequate hepatic function as evidenced by a total bilirubin of <1.5 x upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2) at the time vaccination commences.

Design:

* Following recovery from standard combined modality therapy, patients with no evidence of disease or minimal residual disease will be vaccinated via subcutaneous intradermal injection with 1x10(8) irradiated K562-GM-tumor cells periodically over 6 months. Sterility, potency and identity of the vaccines preps will be confirmed before administration.
* Vaccines will be administered in conjunction with metronomic oral cyclophosphamide and celecoxib.
* Systemic toxicities, and immunologic response to therapy will be recorded. Pre and post vaccination serologic responses to a standard panel of CT antigens as well as cell mediated responses to epigenetically-modified autologous EBV-transformed B and autologous tumor cells (if available) will be assessed before and after vaccination.
* Numbers/percentages and function of T regulatory cells in peripheral blood will be assessed before, during, and after vaccinations.
* Patients will be followed in the clinic with routine staging scans until disease recurrence.
* As the exact set of comparisons and analyses to be performed will be determined following completion of the trial, and will be based on limited numbers of patients, the analyses will be considered exploratory and hypothesis generating rather than definitive.
* Approximately 25 patients will be accrued to this trial.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients with primary small cell or non-small cell lung cancer, esophageal cancer, thymoma, thymic carcinoma, primary sarcoma of the chest, or pleural mesothelioma with no evidence of disease (NED) or minimal residual disease (MRD) in the primary site following standard multi-modality therapy.
2. Patients must be evaluated within 52 weeks following completion of standard therapy and have shown no evidence of disease during that time.
3. Patients with intracranial metastases, which have been treated by surgery or radiation therapy may be eligible for study provided there is no evidence of active disease and no requirement for anticonvulsant therapy or steroids following treatment.
4. Patients must have an ECOG performance status of 0 - 2.
5. Patients must be 18 years of age or older due to the unknown effects of immunologic responses to germ cell-restricted gene products during childhood and adolescent development.
6. Patients must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters:

   * Absolute neutrophil count greater than 1500/mm^3
   * Platelet count greater than 100,000/mm^3
   * Hemoglobin greater than 8g/dl (patients may receive transfusions to meet this parameter)
   * PT within 2 seconds of the ULN
   * Total bilirubin <1.5 times upper limits of normal
   * Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).
7. Seronegative for HIV antibody. Note: The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus may be less responsive to the experimental treatment.
8. Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
9. Patients must be willing to practice birth control during and for four months following treatment.
10. Patients must be willing to sign an informed consent.
11. Patients must be willing to sign an informed consent.

EXCLUSION CRITERIA:

1. Patients who are initially rendered NED or MRD by combined modality therapy but exhibit disease progression prior to initiation of vaccination will be excluded from the study.
2. Patients who will have received more than two systemic cytotoxic treatment regimens for their thoracic malignancy by the time vaccination commences will be excluded.
3. Patients requiring corticosteroids (other than inhaled) will be excluded.
4. Patients with life expectancy less than 12 months will be excluded.
5. Patients receiving warfarin anticoagulation, who cannot be transferred to other agents such as enoxaparin or dabigatran, and for whom anticoagulants cannot be held for up to 24 hours will be excluded.
6. Patients with uncontrolled hypertension (>160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated CHF (>NYHA Class II), or myocardial infarction within 6 months of study will be excluded.
7. Patients with other cardiac diseases may be excluded at the discretion of the PI following consultation with Cardiology consultants.
8. Patients with any of the following pulmonary function abnormalities will be excluded: FEV, < 30% predicted; DLCO < 30% predicted (post-bronchodilator); Oxygen Saturation less than 90% on room air.
9. Pregnant and/or lactating women will be excluded due to the unknown, potentially harmful effects of immune response to CT-X antigens and stem cell proteins that may be expressed in placenta, fetus, and neonates.
10. Patients with active infections, including HIV, will be excluded, due to unknown effects of the vaccine on lymphoid precursors.
11. Patients with any type of primary immunodeficiencies will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-12-07 (Actual); Primary Completion 2015-02-09 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Tabulation of toxicity type and grade | 2 years
  If 25 patients are enrolled and the true probability of a grade 3 or worse toxicity (of any sort) were 20%, then the probability of having 4 or more patients with this occurring is 76.6%. On the other hand, if the combination was very safe and the true probability of a grade 3 or worse toxicity was 5%, then the probability of having 4 or more patients with this occurring would be 3.4%. Thus, if 25 patients were treated, the combination may be considered to have potentially lower safety than tolerable if 4 or more patients experience grade 3 or worse toxicity.

SECONDARY OUTCOMES:
To ascertain if K526-GM vaccines induce immunity to CT antigens commonly expressed in thoracic malignancies. | 2 years
  Perform exploratory analyses which investigate immunologic responses to a panel of CT antigens in vaccinated patients.
To determine if metronomic oral CP and celecoxib reduce the number, percentage and function of CD4+ CD25+ Fox P3+ regulatory T cells (T reg) in peripheral blood of thoracic oncology patients. | 2 years
  Measure T regulatory cells at baseline and at the conclusion of treatment. The difference, or the relative difference, in the values at the two time points will be obtained, and tested to determine if the difference is equal to zero. If a paired t-test is able to be used, with at least 20 evaluable patients, there is 81% power to detect a change equal to 3/4ths of a standard deviation of the change at the two-sided 0.025 significance level.

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kelsen DP, Winter KA, Gunderson LL, Mortimer J, Estes NC, Haller DG, Ajani JA, Kocha W, Minsky BD, Roth JA, Willett CG; Radiation Therapy Oncology Group; USA Intergroup. Long-term results of RTOG trial 8911 (USA Intergroup 113): a random assignment trial comparison of chemotherapy followed by surgery compared with surgery alone for esophageal cancer. J Clin Oncol. 2007 Aug 20;25(24):3719-25. doi: 10.1200/JCO.2006.10.4760. PMID 17704421
- [Background] Manegold C, Thatcher N. Survival improvement in thoracic cancer: progress from the last decade and beyond. Lung Cancer. 2007 Aug;57 Suppl 2:S3-5. doi: 10.1016/S0169-5002(07)70420-8. PMID 17686443
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0138.html